CLINICAL TRIAL: NCT07029295
Title: Evaluation of the Impact of a Patient Education Protocol on the Quality of 18F-FDG PET Imaging Indicated for Investigation of Cardiac Inflammation
Acronym: CARTEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: APHP250343; 2025-A00410-49 (Other: French national Agency for the Safety of Medicines and Health Products); 25.00839.000457 (Other: Commission Nationale des Recherches Impliquant la Personne Humaine)
Record Dates: First submitted 2025-05-27; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Infective Endocarditis; Cardiac Sarcoidosis
Keywords: 18F-FDG; PET; infective endocarditis; cardiac sarcoidosis; patient preparation; patient education protocol
MeSH Terms: conditions — Endocarditis | interventions — 3-Hydroxybutyric Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in two parallel groups:
  * Control group: standard procedure (transmission of instructions sent by e-mail) + compliance questionnaire to be completed on arrival in the day of imaging + BHB (Beta-hydroxybutyrate) assay on capillary blood before imaging.
  * Intervention group: standard procedure accompanied by a link to the educational video (3 min, 34 sec.) prepared as part of the study, explaining the importance of proper preparation and the diet to follow + compliance questionnaire to be completed on arrival in the day of imaging + BHB assay on capillary blood prior to imaging.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): standard procedure (transmission of an instructions sent by e-mail) + compliance questionnaire to be completed on arrival in the day of imaging + BHB assay on capillary blood before imaging.
  Interventions: Behavioral: Compliance questionnaire; Biological: Determination of beta-hydroxybutyrate (BHB) in capillary blood
- Intervention group (Experimental): standard procedure accompanied by a link to the educational video (3 min, 34 sec.) prepared as part of the study, explaining the importance of proper preparation and the diet to follow + compliance questionnaire to be completed on arrival in the day of imaging + BHB assay on capillary blood prior to imaging.
  Interventions: Other: Sending a link to the video; Behavioral: Compliance questionnaire; Biological: Determination of beta-hydroxybutyrate (BHB) in capillary blood

INTERVENTIONS:
Other: Sending a link to the video — Sending a link to the educational video (3 min, 34 sec.) prepared as part of the study, explaining the importance of proper preparation and the diet to follow.
  Arms: Intervention group
Behavioral: Compliance questionnaire — Patient completes a questionnaire on compliance with preparation instructions on the day of the imaging test.
Biological: Determination of beta-hydroxybutyrate (BHB) in capillary blood — Determination of beta-hydroxybutyrate (BHB) in capillary blood prior to imaging examination.

SUMMARY:
The aim of this study is to assess the impact of implementing a patient education and preparation protocol for FDG PET (18F-FDG PET) imaging on the quality of imaging results.

18F-FDG (18Fluor-FluoroDesoxyGlucose) PET (Positron Emission Tomography) is indicated for the diagnosis of cardiac inflammation. To detect cardiac inflammation, the myocardium (heart muscle) must be prevented from absorbing glucose from the diet (FDG). To achieve this, patient preparation is essential. Poor preparation can compromise the interpretation of results, causing diagnostic delay.

To answer the research question, the investigators plan to include 138 people with suspected infective endocarditis or cardiac sarcoidosis, in two institutions of the Assistance Publique - Hôpitaux de Paris: Hôpital Européen Georges Pompidou and Hôpital Cochin-Port-Royal, located respectively at 20 rue Leblanc 75015 Paris and 27 rue du Faubourg Saint-Jacques 75014 Paris.

DETAILED DESCRIPTION:
18F-FDG (18Fluor-FluoroDesoxyGlucose) PET (Positron Emission Tomography) is indicated for the diagnosis of infective endocarditis or cardiac sarcoidosis. Detection of cardiac inflammation requires suppression of physiological glucose (FDG) uptake in the myocardium. To achieve this, patient preparation (ketogenic diet and fasting) is essential. Failure rates vary from center to center. Poor preparation can compromise interpretation, causing diagnostic delay, additional exposure to ionizing radiation and cost. Interpretation of the examination requires suppressing FDG uptake in the myocardium in order to identify FDG uptake in activated inflammatory cells. With this study, the investigators hope to demonstrate that an intervention upstream of the examination will increase the success rate of the 18F-FDG PET examination indicated for cardiac sarcoidosis or infective endocarditis. This will make it possible to avoid reprogramming the examination in the event of failure, and thus limit the patient's additional exposure to ionizing radiation (radiation protection), and avoid a loss of chance for the patient as well as additional costs for health insurance.

Main objective: To evaluate the benefit of implementing a patient education protocol prior to myocardial 18F-FDG PET on the removal of residual myocardial fixation compared with the usual procedure of sending instructions.

Primary endpoint: Success rate of suppression of residual myocardial FDG uptake. Success criteria according to 4 grades. Grade 1 (no residual FDG fixation), grade 2 (moderate FDG fixation in basal LV segments), grade 3 (residual FDG fixation interfering with interpretation) or grade 4 (diffuse and intense FDG fixation). Grades 1 and 2 define success.

Secondary objectives: By comparing the control group (usual procedure) with the intervention group (new procedure):

A - Evaluate the value of determining ketone bodies in capillary blood before the 18F-FDG PET examination indicated for infectious endocarditis or cardiac sarcoidosis, to predict its success.

B - Evaluate whether the patient education protocol leads to greater compliance with dietary instructions prior to the 18F-FDG PET scan.

C - Investigate whether certain drug excipients are likely to influence the results of the 18F-FDG PET scan, by retrieving the list of drugs taken by the patient 24 hours prior to the scan. Indeed, some excipients may contain fast sugars and this could, perhaps, independently of compliance with dietary instructions, lead to failure of the 18F-FDG PET scan.

Secondary endpoints:

A - Measurement of ketone bodies (BHB) on a capillary blood sample taken just before the examination.

B - Use of a questionnaire (cf. appendix 2) drawn up and distributed by the radio handlers to the patient on arrival in the department on the day of the examination.

C - Collection of medications taken by the patient in the 24 hours preceding the examination.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a prescription validated by the nuclear medicine department for an 18F-FDG PET scan for the detection of inflammation of cardiac inflammation or infection
* Age greater than or equal to 18
* Membership of a social security scheme or equivalent
* Patients with an e-mail address
* Patients who understand French
* Collection of patient consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Patients (inpatients or outpatients) already on a diet (including ketogenic)
* Patients who do not understand protocol
* Patients deprived of liberty by judicial or administrative decision
* Patients under legal protection (guardianship/trusteeship)
* Patients under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the benefit of implementing a patient education protocol prior to myocardial 18F-FDG PET on the removal of residual myocardial fixation compared to the usual procedure of sending instructions. | After the imaging (approximately 1 month after the appointment is scheduled for the imaging)
  Interpretation of imaging results :
  Success rate of suppression of residual myocardial FDG uptake. Success criteria according to 4 grades. Grade 1 (no residual FDG uptake), grade 2 (moderate FDG uptake in basal LV segments), grade 3 (residual FDG fixation interfering with interpretation) or grade 4 (diffuse, intense FDG uptake). Grades 1 and 2 define success.
  Centralized review by two independent nuclear medicine physicians and definition of residual FDG uptake in the myocardium blinded to the inclusion group. If there was a discrepancy between the scores, rereading by a 3rd nuclear physician.

SECONDARY OUTCOMES:
Evaluate the value of determining ketone bodies in capillary blood prior to the 18F-FDG PET indicated for infectious endocarditis or cardiac sarcoidosis to predict its success | Before the imaging (approximately 1 month after the appointment is scheduled for the imaging)
  Measurement of ketone bodies (BHB) on a capillary blood sample just before the imaging.
Evaluate whether the patient education protocol leads to greater compliance with dietary instructions prior to 18F-FDG PET. | Before the imaging (approximately 1 month after the appointment is scheduled for the imaging)
  Use of a questionnaire prepared and distributed by radio operators to the patient on arrival on the day of the imaging.
Investigate whether certain drug excipients are likely to influence PET-18F-FDG results | Before the imaging (approximately 1 month after the appointment is scheduled for the imaging)
  Collection of medications taken by the patient in the 24 hours preceding the imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Julien HO, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Cochin - AP-HP, Service de médecine nucléaire, Paris
  - Hôpital Européen Georges Pompidou - AP-HP, Service de médecine nucléaire, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).